CLINICAL TRIAL: NCT04655989
Title: A Prospective, Multi-Center, Randomized, Controlled Trial to Demonstrate the Safety and Effectiveness of the NIKKISO DBB-EXA ES Hemodialysis Delivery System in Adult Patients With Chronic Renal Failure
Brief Title: A Study to Demonstrate the Safety and Effectiveness of the NIKKISO DBB-EXA ES Hemodialysis Delivery System
Acronym: HEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nikkiso America, Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Principal Investigator, Robert Provenzano, MD, Consultant -Office of Chief Medical Officer, Nikkiso America, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DBB-EXA ES-001
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Dialysis; Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Group A subjects will be assigned to 4 weeks of routine dialysis (control group) followed by 4 weeks of treatment dialysis with the DBB-EXA ES Hemodialysis System (investigational group).
  Group B subjects will be assigned to 4 weeks of treatment dialysis with the DBB-EXA ES Hemodialysis System (investigational group) followed by 4 weeks of routine dialysis (control group).
  After completion of the initial 8-week treatment period, subjects were eligible for the Vascular Access Recirculation Rate Measurement (VARRM) sub-study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Routine first (Experimental): Group A subjects will be assigned to 4 weeks of routine dialysis (control group) followed by 4 weeks of treatment dialysis with the DBB-EXA ES Hemodialysis System (investigational group).
  Interventions: Device: DBB-EXA ES Hemodialysis System
- Investigational first (Experimental): Group B subjects will be assigned to 4 weeks of treatment dialysis with the DBB-EXA ES Hemodialysis System (investigational group) followed by 4 weeks of routine dialysis (control group).
  Interventions: Device: DBB-EXA ES Hemodialysis System
- VARRM sub-study (Other): Following completion of the initial 8-week treatment, subject's were eligible to participate in the sub-study, VARRM. The total participation time for the VARRM sub-study was approximately 1.5 weeks.
  Interventions: Device: DBB-EXA ES Hemodialysis System

INTERVENTIONS:
Device: DBB-EXA ES Hemodialysis System — The DBB-EXA ES Hemodialysis Delivery System is intended to support an optional online priming, rinseback and emergency bolus features. The appropriate priming of the hollow fiber dialyzer and blood tubing lines removes debris and air prior to device use, as well as ensuring proper rinseback.

SUMMARY:
The study objective is to verify the safety and effectiveness of the DBB-EXA ES Hemodialysis Delivery System to consistently deliver dialysate of the appropriate quality for infusion.

DETAILED DESCRIPTION:
The study objective is to verify the safety and effectiveness of the DBB-EXA ES Hemodialysis Delivery System to consistently deliver dialysate of the appropriate quality for infusion. The safety will be evaluated by comparing the adverse event rate in the DBB-EXA ES Hemodialysis group (investigational) vs. the standard dialysis group (control).

The study population will include eligible adult patients diagnosed with chronic renal failure requiring routine dialysis treatments for a minimum of 90 days and with a minimum of 3 weekly sessions. Treatment duration will be at the discretion of the investigator. The duration of study participation for each subject is approximately eight (8) weeks; four (4) weeks of routine dialysis and four (4) weeks of treatment dialysis. The expected total study duration across all subjects (from recruitment to last subject visits) is approximately five (5) to six (6) months, dependent upon subject recruitment/enrollment and meeting 360 evaluable treatments. A minimum of 30 eligible subjects will be enrolled into the study ensuring a minimum of 360 evaluable treatments in the treatment arm.

The sub-study, VARRM, was conducted following the subject's completion of the primary eight (8) week clinical study. The total participation time for the VARRM sub-study was approximately 1.5 weeks. Subjects that participated in the VARRM sub-study had their vascular recirculation rates collected during treatments. A minimum of 12 subjects were expected to participate in this sub-study, with a minimum of 21 and maximum of 36 dialysis accesses evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Chronic renal failure diagnosis
3. Minimum of 90 days of stable hemodialysis treatment with a minimum of 3 treatment sessions per week. The duration of each treatment session is in the discretion of the investigator.
4. Reliable vascular access
5. Hemodialysis treatment a minimum of three (3) sessions per week
6. Subject agrees not to eat or drink during treatments
7. Understand and sign the informed consent form

Exclusion Criteria:

1. Unable to receive anticoagulation
2. Hypercoagulation diagnosis
3. Hyperviscosity diagnosis
4. Most recent hemoglobin less than 9
5. Active bacterial infection
6. Women of childbearing potential, pregnant and/or lactating females verified by urine or serum pregnancy test
7. Life expectancy less than 6 months
8. Cognitive impairment, dementia, or other condition that limits the ability to provide informed consent and to comply with study procedures, or any other reason that the Investigator believes to contraindicate study participation.
9. Current or known future need for a central venous catheter (CVC)
10. Involved in another clinical research trial within the prior 30 days
11. Diagnosed with systemic consistent hypotension as defined by being systolic <90 mm Hg or diastolic <60 mm Hg
12. Immunocompromised patients (e.g. active malignancy, current chemotherapy treatment, transplant recipients, any patient on immunosuppressive medication, or patients with current autoimmune disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Adverse Event Rate | 8 weeks
  The safety will be evaluated by comparing the adverse event rate in the DBB-EXA ES Hemodialysis group (investigational) vs. the standard dialysis group (control)

SECONDARY OUTCOMES:
Total Colony Forming Units and Endotoxin Levels | 8 Weeks
  The effectiveness will be evaluated by comparing the total Colony Forming Units (CFUs) and endotoxin levels calculated within dialysis fluid in the DBB-EXA ES Hemodialysis group (investigational) vs. the standard dialysis group (control).
Fluid Balance Evaluation | 8 Weeks
  The impact that online priming, online rinse back and online emergency bolus, if performed, has on fluid balance will be evaluated by assessing the proportion of subjects that have a Post-Dialysis Target Weight variance of > 0.5kg in the DBB-EXA ES Hemodialysis group (investigational) vs. the standard dialysis group (control).

OTHER OUTCOMES:
Sub-Study VARRM | 1.5 weeks
  The Vascular Access Recirculation Rate Measurement (VARRM) will be assessed by comparing the recirculation rate obtained from the DBB-EXA ES device to the non-invasive commercially approved Transonic® HD03 Hemodialysis Monitor (Transonic Systems, Inc.)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Great Lakes Dialysis, Detroit, Michigan
  - Great Lakes Dialysis - West, Southfield, Michigan

IPD SHARING:
Plan to Share IPD: No